CLINICAL TRIAL: NCT01206764
Title: An Open-label, Multi-center Phase 2 Study to Evaluate Everolimus as Monotherapy Treatment for Patients With Metastatic Recurrent and/or Unresectable Renal Cell Carcinoma (EVERMORE).
Brief Title: A Trial of Everolimis in Patients With Advanced Renal Cell Carcinoma.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001LIC01
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC,; mTOR pathway,; angiogenesis,; PFS,; partial response [PR] + complete response [CR]); metastatic recurrent renal cell carcinoma; metastatic unresectable renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAD001 (Experimental)
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001
  Other Names: Everolimus

SUMMARY:
Renal cell carcinoma (RCC) accounts for more than 200,000 new cases of cancer and over 100,000 cancer deaths annually in the World (Ferlay, et al., 2004). It is estimated that there were about 15,000 new cases of RCC in the region that excludes the Americas, European Union and Japan. Renal cell carcinomas arise from the proximal tubal epithelium are more common in males than in females with an overall lifetime risk of 1 in 75 and a median age of diagnosis of 65 years.

Everolimus (Certican®) has been approved since 2003 in more than 60 countries for the prevention of organ rejection in patients with renal and cardiac transplantation. Everolimus (RAD001) is a derivative of rapamycin, which acts as a signal transduction inhibitor. It targets mTOR, a key protein kinase regulating cell growth, proliferation, and survival. The mTOR pathway activity is modulated by the phosphatidylinositol-3-kinase (PI3K)/protein kinase B AKT (AKT) pathway, a pathway known to be deregulated in numerous human cancers. RAD001 (Afinitor®) has been investigated as an anticancer agent based on its potential to act:

* directly on the tumor cells by inhibiting tumor cell growth and proliferation;
* indirectly by inhibiting angiogenesis leading to reduced tumor vascularity (via potent inhibition of tumor cell hypoxia-inducible factor 1 (HIF-1) activity, VEGF production, and VEGF-induced proliferation of endothelial cells).

Primary: To evaluate the PFS rate over time.

Secondary:

* To evaluate the disease control rate (stable disease [SD] + partial response [PR] + complete response [CR]);
* To evaluate the objective response rate (ORR; where ORR = CR + PR) and duration;
* To describe the safety profile of RAD001.

ELIGIBILITY:
Inclusion Criteria: Patients may be entered in the study only if they meet all of the following criteria:

* Age ≥18 years old;
* Patients with advanced renal cell carcinoma with confirmed clear or non-clear cell histology, with or without nephrectomy, and with any MSKCC prognosis;
* Prior cytokine therapy is permitted;
* Patients with at least one measurable lesion at baseline as per the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. If skin lesions are reported as target lesions, they must be documented (at baseline and at every physical exam) using color photography and a measuring device (such as a caliper) in clear focus to allow the size of the lesion(s) to be determined from the photograph;
* Life expectancy ≥3 months. Life expectancy should be judged in relation to other determining patient eligibility factors such as laboratory results, Karnofsky Performance Status, etc.;
* Patients with a Karnofsky Performance Status ≥70%;
* Adequate bone marrow function as shown by: absolute neutrophil count (ANC) ≥1.5 x 109/L, platelets ≥100 x 109/L, hemoglobin (Hb) >9 g/dL;
* Adequate liver function: serum bilirubin ≤1.5 x upper limit of normal (ULN), alanine transaminase (ALT), and aspartate transaminase (AST) ≤2.5 x ULN;
* Adequate renal function: serum creatinine ≤1.5 x ULN;
* Females of childbearing potential must have had a negative serum or urine pregnancy test 7 days prior to the administration of the study treatment start;
* Patients who give a written informed consent obtained according to local guidelines.

Exclusion Criteria:Patients may not be entered into the study if they meet any of the following criteria:

* Patients within 2 weeks post-minor surgery (e.g., herniorrhaphy), 4 weeks post-major surgery (e.g., intra-thoracic, intra-abdominal, or intra-pelvic) to avoid wound healing complications. Percutaneous biopsies require no waiting time prior to study entry;
* Patients with a recent history of hemoptysis, ≥0.5 teaspoon of red blood;
* Patients who have received prior systemic treatment for their metastatic RCC other than with cytokine therapy;
* Patients who received prior therapy with a VEGF pathway inhibitor, such as sunitinib, sorafenib, and bevacizumab;
* Patients who have previously received mTOR inhibitors (sirolimus, temsirolimus, everolimus, deferolimus);
* History or clinical evidence of central nervous system (CNS) metastases. Note: Subjects who have previously-treated CNS metastases (surgery ± radiotherapy, radiosurgery, or gamma knife) and meet all 3 of the following criteria are eligible:

Are asymptomatic; Have had no evidence of active CNS metastases for ≥6 months prior to enrollment and; Have no requirement for steroids or enzyme-inducing anticonvulsants (EIAC);

• Clinically significant gastrointestinal abnormalities including, but not limited to: Malabsorption syndrome; Major resection of the stomach or small bowel that could affect the absorption of study drug; Active peptic ulcer disease; Inflammatory bowel disease; Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation; History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning of study treatment;

* Patients receiving chronic systemic treatment with corticosteroids (dose of ≥10 mg/day methylprednisone equivalent) or another immune-suppressive agent. Inhaled and topical steroids are acceptable, as well as opotherapy after bilateral adrenal gland removal;
* Patients with a known history of human immunodeficiency virus seropositivity;
* Patients with autoimmune hepatitis;
* Patients with an active, bleeding diathesis. Patients may use coumadin or heparin preparations;
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study;
* Patients who have a history of another primary malignancy ≤3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of uterine;
* Female patients who are pregnant or breastfeeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the study by both sexes. Oral contraceptives are not acceptable;
* Patients who are using other investigational agents or who had received investigational drugs ≤4 weeks prior to study treatment start; Patients unwilling or unable to comply with the protocol.

Other protocol-defined inclusion/exclusion may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-11-11 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Algeria (2):
  - Novartis Investigative Site, Algiers
  - Novartis Investigative Site, Oran
- Egypt (3):
  - Novartis Investigative Site, Al Mansurah
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- India (2):
  - Novartis Investigative Site, Indore, Madhya Pradesh
  - Novartis Investigative Site, Pune, Maharashtra
- Novartis Investigative Site, Amman, Jordan
- Novartis Investigative Site, El Achrafiyé, Lebanon
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Samara
- Novartis Investigative Site, Riyadh, Saudi Arabia
- South Africa (3):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Parktown
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Tunisia (3):
  - Novartis Investigative Site, Tunis, Tunisie
  - Novartis Investigative Site, Aryanah
  - Novartis Investigative Site, Sousse

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001: Two 5 mg RAD001 tablets
Period: Overall Study
Arm/Group | RAD001
Started | 142
Completed | 4
Not Completed | 138
Not completed — Adverse Event | 20
Not completed — Abnormal laboratory value | 2
Not completed — Abnormal test procedure result | 1
Not completed — Patient withdrew consent | 5
Not completed — Lost to Follow-up | 6
Not completed — Death | 11
Not completed — New cancer therapy | 2
Not completed — Disease progression | 88
Not completed — Protocol deviation | 3

BASELINE CHARACTERISTICS:
Arm/Group | RAD001
Number analyzed (Participants) | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 42
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 71
  More than one race | 0
  Unknown or Not Reported | 27

OUTCOME MEASURES:

1. Primary Outcome: PFS (Progression-Free Survival)
Description: the time from the date of the start of RAD001 treatment to the date of the first documented disease progression or death due to any cause
Time Frame: Approximately 4 years
Population: The Intent-to-Treat population (ITT population) consisted of all patients treated with RAD001.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | RAD001
Number analyzed (Participants) | 142
Weeks | 27.71 [21.86 to 35.29]
Statistical Analysis 1: Comparison: RAD001; Single arm open label study; Test type: Other — Kaplan Meier; Median Difference (Net) = 27.71, 95% CI 2-sided [21.86 to 35.29]

2. Secondary Outcome: Disease Control Rate (Stable Disease [SD] + Partial Response [PR] + Complete Response [CR]);
Description: The disease control rate was based on the data as per local radiological review following the RECIST criteria. The disease control rate is defined as the proportion of patients with CR, PR, or SD and was summarized in terms of percentage with 95% exact Clopper-Pearson CIs
Time Frame: Approximately 4 years
Population: The Intent-to-Treat population (ITT population) consisted of all patients treated with RAD001.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | RAD001
Number analyzed (Participants) | 142
Percentage of Participants | 74.6 [66.7 to 81.6]

3. Secondary Outcome: Objective Response Rate (ORR; Where ORR = CR + PR)
Description: The overall tumor response was based on the data as per local radiological review, following RECIST criteria. The ORR is defined as the proportion of patients with CR or PR and was summarized in terms of percentage with 95% exact Clopper-Pearson CIs
Time Frame: Approximately 4 years
Population: The Intent-to-Treat population (ITT population) consisted of all patients treated with RAD001.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RAD001
Number analyzed (Participants) | 142
Percentage of participants | 17 [7.1 to 18.5]

4. Secondary Outcome: Duration of Response (DOR)
Description: The DOR analysis applied only to patients whose overall response was CR or PR and was defined as the time from onset of response (CR/PR) to progression or death from any cause
Time Frame: Approximately 4 years
Population: The Intent-to-Treat population (ITT population) consisted of all patients treated with RAD001.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | RAD001
Number analyzed (Participants) | 142
Weeks | 169 [52.71 to NA] — NA= level of detection, insufficient number of participants with events

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of start of treatment to date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last contact.
Time Frame: Approximately 4 years
Population: The Intent-to-Treat population (ITT population) consisted of all patients treated with RAD001.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | RAD001
Number analyzed (Participants) | 142
Weeks | NA [116.86 to NA] — NA=level of detection, insufficient number of participants with events
Statistical Analysis 1: Comparison: RAD001; The median overall survival was not evaluable, this presents the 25th percentile of overall survival; Test type: Other — Kaplan Meier; Median Difference (Net) = 45.71, 95% CI 2-sided [31.29 to 106.43]

ADVERSE EVENTS:
Time Frame: Approximately 4 years
Description: AE additional description
Arm/Group | RAD001
All-Cause Mortality (participants affected / at risk) | 33/142
Serious Adverse Events (participants affected / at risk) | 48/142
Other Adverse Events (participants affected / at risk) | 125/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=142)
ANAEMIA (Blood and lymphatic system disorders) | 5
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 1
HYPERCALCAEMIA OF MALIGNANCY (Endocrine disorders) | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
COLONIC FISTULA (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 3
DYSPHAGIA (Gastrointestinal disorders) | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 2
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 3
FATIGUE (General disorders) | 1
MUCOSAL INFLAMMATION (General disorders) | 4
MULTI-ORGAN DISORDER (General disorders) | 1
PYREXIA (General disorders) | 1
ABSCESS (Infections and infestations) | 1
ANAL ABSCESS (Infections and infestations) | 1
BACTERAEMIA (Infections and infestations) | 1
DIVERTICULITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
GENITAL ABSCESS (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 6
SEPSIS (Infections and infestations) | 2
TOOTH ABSCESS (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 3
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
BLOOD CREATININE INCREASED (Investigations) | 2
URINE OUTPUT DECREASED (Investigations) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
DEHYDRATION (Metabolism and nutrition disorders) | 3
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1
KETOACIDOSIS (Metabolism and nutrition disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
BONE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1
HEMIPARESIS (Nervous system disorders) | 2
LETHARGY (Nervous system disorders) | 1
MENTAL IMPAIRMENT (Nervous system disorders) | 1
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
HAEMATURIA (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3
RENAL IMPAIRMENT (Renal and urinary disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1
HYPOTENSION (Vascular disorders) | 1
THROMBOPHLEBITIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=142)
ANAEMIA (Blood and lymphatic system disorders) | 62
LEUKOPENIA (Blood and lymphatic system disorders) | 22
NEUTROPENIA (Blood and lymphatic system disorders) | 23
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 18
ABDOMINAL PAIN (Gastrointestinal disorders) | 15
CONSTIPATION (Gastrointestinal disorders) | 15
DIARRHOEA (Gastrointestinal disorders) | 18
NAUSEA (Gastrointestinal disorders) | 15
STOMATITIS (Gastrointestinal disorders) | 41
VOMITING (Gastrointestinal disorders) | 9
ASTHENIA (General disorders) | 22
FATIGUE (General disorders) | 30
MUCOSAL INFLAMMATION (General disorders) | 24
OEDEMA PERIPHERAL (General disorders) | 15
PYREXIA (General disorders) | 14
URINARY TRACT INFECTION (Infections and infestations) | 9
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 14
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 16
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 11
BLOOD CHOLESTEROL INCREASED (Investigations) | 13
BLOOD CREATININE INCREASED (Investigations) | 21
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 12
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 19
PROTHROMBIN TIME PROLONGED (Investigations) | 8
ABNORMAL LOSS OF WEIGHT (Metabolism and nutrition disorders) | 29
DECREASED APPETITE (Metabolism and nutrition disorders) | 32
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 25
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 37
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 10
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 21
HYPERURICAEMIA (Metabolism and nutrition disorders) | 10
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 11
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 18
HYPOKALAEMIA (Metabolism and nutrition disorders) | 9
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 12
DYSGEUSIA (Nervous system disorders) | 9
HEADACHE (Nervous system disorders) | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 31
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 20
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 16
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 11
PRURITUS (Skin and subcutaneous tissue disorders) | 11
RASH (Skin and subcutaneous tissue disorders) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT01206764/SAP_000.pdf
  • Study Protocol (2010-05-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT01206764/Prot_001.pdf